CLINICAL TRIAL: NCT03420495
Title: Decision-making Impairments in OCD: An Integrated Behavioral Economics Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Obsessive Compulsive Foundation (Other)
Responsible Party: Principal Investigator, Ryan Jane Jacoby, Ryan Jane Jacoby, Ph.D., Clinical Psychologist, OCD and Related Disorders Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P002668
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Intolerance of Uncertainty
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The current study has two diagnostic arms (the OCD group and the Non-Psychiatric Control group) all receiving a single interventional protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCD Group (Experimental): Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for principal OCD. These participants will complete clinician interviews, self-report questionnaires, and receive the Decision-Making Tasks Intervention.
  Interventions: Behavioral: Decision-Making Tasks
- Non-psychiatric Control Group (Experimental): No current DSM-5 diagnosis. These participants will also complete clinician interviews, self-report questionnaires, and receive the Decision-Making Tasks Intervention.
  Interventions: Behavioral: Decision-Making Tasks

INTERVENTIONS:
Behavioral: Decision-Making Tasks — All participants will receive a structured diagnostic assessment and complete self-report questionnaires about cognitive factors, decision-making styles, and anxiety/mood symptoms. They then will be guided through three judgment and decision-making (JDM) paradigms (the Risk and Ambiguity Task, the Beads Task, and the Balloon Analogue Risk Task), each of which each has been modified to differ by whether the likelihood of potential adverse outcomes is provided (or whether it remains ambiguous).

SUMMARY:
The investigators are examining whether conditions of ambiguity during decision-making may prime intolerance of uncertainty beliefs (i.e., difficulties coping with ambiguity, unpredictability, and the future) and lead to impaired performance when individuals with obsessive-compulsive disorder (OCD) are making uncertain decisions compared to non-psychiatric controls.

DETAILED DESCRIPTION:
The primary aims of this study are to examine the extent to which individuals with OCD avoid decisions that involve ambiguity through the use of self-report and behavioral measures. Specifically, the investigators will examine how individuals with OCD minimize risk at the expense of monetary profit under conditions of ambiguity (relative to risky but unambiguous options) compared to non-psychiatric controls utilizing a series of judgment and decision-making (JDM) tasks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18+)
* Meet DSM-5 criteria for principal OCD (OCD group) or no current DSM-5 diagnosis (NPC group).
* Sufficient fluency of English to understand study procedures and questionnaires
* Ability to provide informed consent.
* Comfortable and capable of using a computer to complete computer-based decision-making tasks.

Exclusion Criteria:

* Color-blindness (which prevents completion of certain tasks)
* Acute psychosis, bipolar disorder, substance use disorder, or suicidality. All other diagnostic comorbidities will be permitted to foster the accrual of a clinically relevant sample.
* Serious neurological disorder or impairment (e.g., brain damage, blindness), attention deficit hyperactivity disorder (ADHD), intellectual disability, or autism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Ambiguity aversion score on the Risk and Ambiguity Task | Day 1
  In the Risk and Ambiguity Task participants make repeated choices between a certain payoff vs. a gamble. On low ambiguity trials, the likelihood of the gamble is known (i.e., "risky" lottery). On high ambiguity trials, the likelihood of the gamble is unknown (i.e., "ambiguous" lottery). Ambiguity aversion = (number of 50% risky lotteries chosen / total number of 50% risky lotteries) - (# of ambiguous lotteries chosen / total number of ambiguous lotteries).
Average adjusted pump scores on the Balloon Analogue Risk Task (BART) | Day 1
  In the BART participants blow up a series of virtual balloons. With each pump: (a) they earn 5 cents that accumulate in a temporary reserve, but (b) the likelihood of the balloon exploding increases. When this occurs participants lose the money in their temporary reserve. At any time, participants can choose to transfer their earnings to a permanent savings bank (and move to the next balloon). Thus, participants weigh the likelihood of the negative outcome (i.e., the balloon exploding and losing money) with the potential gains (i.e., 5 cents per pump). In the low ambiguity version of the task, the likelihood of the balloon exploding is known. In the high ambiguity version, the likelihood of the balloon exploding is unknown. The average adjusted pump score = average number of pumps on trials in which the balloons did not explode.

SECONDARY OUTCOMES:
Money spent on draws to decision (DTD) in the Beads Task | Day 1
  The Beads Task is a probabilistic inference task in which participants gather as much information (i.e., beads) as they desire before feeling "certain" enough to decide from which jar the beads have come. Participants will start off with a fixed amount of money, and invest money for each bead requested. If they answer correctly, the money earned will be transferred to a savings bank; if incorrect, they lose any earnings from that trial. Thus, participants must consider the tradeoff between the number of beads they choose and their accuracy as they decide. In the low ambiguity version of the task, the ratio of colored beads inside the jar is known. In the high ambiguity version, the ratio of colored beads inside the jar is unknown.
Intolerance of Uncertainty Scale (IUS-12) | Day 1
  The IUS-12 measures reactions to uncertainty, ambiguity, and the future consisting of two subscales: Prospective and Inhibitory IU.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Jacoby, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No